CLINICAL TRIAL: NCT06656611
Title: PAPMOBILE: Mobile Outreach Screening of High-Risk Human Papillomavirus Infection in Women with Limited Access to Health Services in Seine-Saint-Denis (greater Paris Area, France)
Brief Title: Mobile Outreach Screening of High-Risk Human Papillomavirus Infection in Women with Limited Access to Health Services in Seine-Saint-Denis (greater Paris Area, France)
Acronym: PAPMOBILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Hospital Avicenne (Other); National Cancer Institute, France (Other Government); INSERM UMR S 1136 (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IMEA 072
Record Dates: First submitted 2024-07-25; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Women's Health: Cervical Neoplasm
Keywords: HPV; cervical cancer; outreach intervention; vaginal self sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prospective cervical cancer screening intervention (Other): Evaluation of a cervical cancer screening outreach intervention using point-of-care High-Risk HPV (HPV-HR) tests on self-collected vaginal swabs
  Interventions: Other: HPV self sampling

INTERVENTIONS:
Other: HPV self sampling — Selected women will perform a vaginal self-sampling using a swab

SUMMARY:
The study is a prospective cervical cancer screening intervention in the nonclinical setting of a mobile testing unit in a vehicle, using point-of-care HPV PCR tests with self-collected vaginal swabs.

It is designed for women with limited access to healthcare and prevention in underprivileged municipalities in the greater Paris area (Seine-Saint-Denis department, detailed in Annexe 3).

HPV positive participants will receive counseiling and guidance to help them find a healthcare professional to take care of their needs

ELIGIBILITY:
Inclusion Criteria:

* - Women from 30 to 65 years of age presenting to the " Bus Santé " nonclinical testing unit, eligible to cervical cancer screening by an HPV-HR test
* Women affiliated to the French social security or immigrants benefiting from the state medical aid program for undocumented immigrants (Aide Médicale d'Etat). The inclusion of people not affiliated to a social security system is an exception and depends on the decision of the Personal Protection Committee, if it is based on an expected benefit for these people of a nature to justify the foreseeable risk incurred.
* The intervention is designed for vulnerable women with limited access to healthcare, including but not limited to:

  * Women living in shelters and hostels, women living in the streets, in squats, hot-bedding arrangements, emergency social housing;
  * Recent immigrants, documented or undocumented;
  * Young adults from priority neighbourhoods,
  * Isolated or marginalized women
* Free, informed, written consent, signed by the person and the investigator at the latest on the day of inclusion and before any sampling carried out as part of the trial (article L1122-1-1 of the Public Health Code)

The Bus will operate in underprivileged neighbourhoods in the greater Paris area (eastern Seine-Saint-Denis department.

Exclusion Criteria:

* Screened for cervical cancer by a PAP smear in the last 3 years or by an HPV test in the last 5 years,
* Women on their period (haemoglobin inhibits PCRs)
* Pregnancy in the 2nd and 3rd trimesters
* Total hysterectomy; absence of a vagina
* Women under guardianship/tutelage

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Total number and proportion of eligible women (age 30 to 65, unscreened for cervical cancer for 3 to 5 years) who had an HPV PCR test on a self-collected vaginal sample when offered in a nonclinical setting by the Bus Santé de Seine-Saint-Denis | Day 0

SECONDARY OUTCOMES:
Declined to participate: number and why | Day 0
Description of the barriers to cervical cancer screening in the target population | Day 0
Proportion of complete HPV-HR PCRs run onboard the Bus and proportion with same-day results available to the participants | Day 0
Frequency of positive HPV-HR tests and of invalid HPV-HR tests using SCVS samples | Day 0
Description of HPV types in the participant population | Day 0
Comparison of HPV-HR negative and HPV-HR positive participants | Day 0
Proportion of secondary pelvic examination and cervical PAP smears in HPV-positive participants ; in Step 1 (laboratory-based PCR) and Step 2 (PCR aboard the Bus with same-day results) | Day 0
Proportion of Chlamydiae trachomatis and Neisseria gonorrhoea STIs | Day 0
Number and frequency of cytological abnormalities and cervical lesions in participants who had a PAP smear following a positive HPV-HR test ; in Step 1 (laboratory-based PCR) and Step 2 (PCR aboard the Bus with same-day results) | Day 0
Proportion of valid self-collected vaginal swabs (cellular density, valid HPV PCR) | Day 0
Unavailability of point-of-care HPV-HR PCR: number of days and why (reagent shortage, instrument of power failure, environmental conditions, short-staffing…) | Day 0
Reliability of vaginal self-sampling in a nonclinical setting: proportion of valid samples, types of non-conformity | Day 0
Participant satisfaction with point-of-care self-sampling and HPV testing; proportion willing to recommend the intervention to their acquaintance | Day 0
Staff satisfaction by self-questionnary | Day 0
Adverse events; setbacks and adjustments over the study period | From day 0 to the last call (about month 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rahib D. Place de l'auto-prélèvement " à domicile " dans les stratégies de dépistage du VIH et des autres infections sexuellement transmissibles chez les hommes ayant des relations sexuelles avec des hommes en France. 2022; Available at: https://theses.fr/api/v1/document/2022SORUS219
- [Background] Reques L, Rolland C, Lallemand A, Lahmidi N, Aranda-Fernandez E, Lazzarino A, Bottero J, Hamers F, Bergeron C, Haguenoer K, Launoy G, Luhmann N. Comparison of cervical cancer screening by self-sampling papillomavirus test versus pap-smear in underprivileged women in France. BMC Womens Health. 2021 May 26;21(1):221. doi: 10.1186/s12905-021-01356-8. PMID 34039341
- [Background] Pretsch PK, Spees LP, Brewer NT, Hudgens MG, Sanusi B, Rohner E, Miller E, Jackson SL, Barclay L, Carter A, Wheeler SB, Smith JS. Effect of HPV self-collection kits on cervical cancer screening uptake among under-screened women from low-income US backgrounds (MBMT-3): a phase 3, open-label, randomised controlled trial. Lancet Public Health. 2023 Jun;8(6):e411-e421. doi: 10.1016/S2468-2667(23)00076-2. Epub 2023 May 11. PMID 37182529
- [Background] CNR HPV. Trousses de détection des HPV ayant bénéficié d'une validation clinique pour le dépistage du cancer du col de l'utérus. 2023; Available at: https://cnr-hpv.fr/wp-content/uploads/2023/03/Liste-des-trousses-de-detection-et-de-genotypage-des-HPV-validees-par-les-fabricants-de-milieux-v11.pdf.
- [Background] Institut National du Cancer, CNR HPV, France. Référentiel national - Dépistage du cancer du col de l'utérus - cadre et modalités de recours aux autoprélèvements vaginaux. 2022; Available at: https://www.e-cancer.fr/Expertises-et-publications/Catalogue-des-publications/Referentiel-national-Depistage-du-cancer-du-col-de-l-uterus-cadre-et-modalites-de-recours-aux-autoprelevements-vaginaux.
- [Background] Dourgnon P, Jusot F, Sermet C, Silva J. La santé perçue des immigrés en France. 2008; Available at: https://www.irdes.fr/Publications/Qes/Qes133.pdf.